CLINICAL TRIAL: NCT01393067
Title: Comparison of Use of Covered, Self-expandable Metal Stents (cSEMS) and Non-expandable Plastic Stents (NEPS) in Temporary Endoscopic Treatment of Stenosis of the Bilio-biliary Anastomosis After Liver Transplantation
Brief Title: cSEMS vs. NEPS in Stricture of Biliary Anastomosis After Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Jorg Albert, Johann Wolfgang Goethe University Hospitals., Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 148/10
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Stenosis of the Bilio-biliary Anastomosis After Orthotopic Liver Transplantation
Keywords: cSEMS; NEPS; ERCP; biliary stricture; biliary stenosis; liver transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group NEPS (Active Comparator): implantation of multiple non-expandable plastic stents
  Interventions: Device: Non-expandable plastic stent (plastic endoprosthesis)
- group cSEMS (Active Comparator): implantation of a self-expandable metal stent (cSEMS)
  Interventions: Device: Covered self-expandable metal stent (cSEMS)

INTERVENTIONS:
Device: Non-expandable plastic stent (plastic endoprosthesis) — plastic stent (plastic endoprosthesis)
  Other Names: OptiMed, Boston Scientifiv, MTW
  Arms: study group NEPS
Device: Covered self-expandable metal stent (cSEMS) — Removable, covered self-expandable metal stent (cSEMS)
  Other Names: Niti-S biliary stent, fully covered
  Arms: group cSEMS

SUMMARY:
Stenosis at the bilio-biliary anastomosis occurs in up to 30% of patients after orthotopic liver transplantation. This study compares endoscopic treatment with implantation of multiple plastic endoprostheses vs. use of a removable, covered self-expandable metal stent (cSEMS).

DETAILED DESCRIPTION:
This is a multi-center randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* post-OLT stenosis of the bilio-biliary anastomotic

Exclusion Criteria:

* non-anastomotic stricture
* stent implatation technically not feasible

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of interventions (ERCP) to attain resolution of stenosis | up to one year
  Number of interventions (ERC) in study group cSEMS is compared to number of interventions (ERC) in study group NEPS

SECONDARY OUTCOMES:
Occurence and severity of complications related to the endoscopic procedures | up to 2 months after ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Albert, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital and Clinics Department of Internal Medicine I
Locations (4):
- University of Helsinki, Helsinki, Finland
- Germany (2):
  - Klinik für Gastroenterologie und Hepatologie, Medizinische Hochschule Essen, Essen
  - Department of Internal Medicine I, Frankfurt
- University of Milano, Milan, Italy

REFERENCES:
- [Background] Kahaleh M, Behm B, Clarke BW, Brock A, Shami VM, De La Rue SA, Sundaram V, Tokar J, Adams RB, Yeaton P. Temporary placement of covered self-expandable metal stents in benign biliary strictures: a new paradigm? (with video). Gastrointest Endosc. 2008 Mar;67(3):446-54. doi: 10.1016/j.gie.2007.06.057. PMID 18294506
- [Background] Wang AY, Ellen K, Berg CL, Schmitt TM, Kahaleh M. Fully covered self-expandable metallic stents in the management of complex biliary leaks: preliminary data - a case series. Endoscopy. 2009 Sep;41(9):781-6. doi: 10.1055/s-0029-1215050. Epub 2009 Aug 19. PMID 19693751
- [Background] Phillips MS, Bonatti H, Sauer BG, Smith L, Javaid M, Kahaleh M, Schmitt T. Elevated stricture rate following the use of fully covered self-expandable metal biliary stents for biliary leaks following liver transplantation. Endoscopy. 2011 Jun;43(6):512-7. doi: 10.1055/s-0030-1256389. Epub 2011 May 26. PMID 21618151
- [Derived] Tal AO, Finkelmeier F, Filmann N, Kylanpaa L, Udd M, Parzanese I, Cantu P, Dechene A, Penndorf V, Schnitzbauer A, Friedrich-Rust M, Zeuzem S, Albert JG. Multiple plastic stents versus covered metal stent for treatment of anastomotic biliary strictures after liver transplantation: a prospective, randomized, multicenter trial. Gastrointest Endosc. 2017 Dec;86(6):1038-1045. doi: 10.1016/j.gie.2017.03.009. Epub 2017 Mar 14. PMID 28302527